CLINICAL TRIAL: NCT02141178
Title: Does Long-Acting Liposomal Bupivacaine Provide Improved Pain Relief Over Bupivicaine Alone in Carpal Tunnel Release?
Brief Title: Comparison of Bupivacaine and Exparel for Carpal Tunnel Release
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No IRB approval
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: PRO14040418
Record Dates: First submitted 2014-05-12; First posted 2014-05-19 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Pain After Carpal Tunnel Release
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Active Comparator): Patients will received 0.5% Bupivacaine subcutaneously for local anesthesia during surgery
  Interventions: Drug: Bupivacaine
- Exparel (Experimental): Patients will received Exparel subcutaneously for local anesthesia during surgery
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Bupivacaine
  Arms: Bupivacaine
Drug: Exparel
  Arms: Exparel

SUMMARY:
Carpal tunnel syndrome is one of the most common surgeries performed per year in the United States, accounting for over 600,000 surgeries. The procedure is commonly performed under light sedation and local anesthesia. Bupivicaine, a long acting local anesthetic, has been used to allow extended pain relief for 8-10 hours after carpal tunnel release. Exparel, a liposomal bupivicaine formulation, has been documented to provide pain relief for up to 72 hours post-operatively. By decreasing post-operative pain through the use of a long-acting local anesthetic, the use of narcotic pain medications may be decreased and patient satisfaction scores may increase.

The purpose of this study is to prospectively compare bupivicaine and liposomal bupivicaine with respect to post-operative pain control, narcotic usage, and patient satisfaction after carpal tunnel release.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carpal tunnel syndrome undergoing surgery

Exclusion Criteria:

* Non english speaking
* Allergy to bupivacaine or exparel

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain | Starting immediately after surgery and then every 8 hours for 10 days
  Pain will be evaluated using an 11-point ordinal scale (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States